CLINICAL TRIAL: NCT02232880
Title: Treatment of Resistant Hypertension by Prevention of T-Cell Co-Stimulation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: failure to recruit
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121740
Record Dates: First submitted 2014-08-12; First posted 2014-09-05 (Estimated); Results first posted 2016-08-29 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Hypertension
Keywords: hypertension; inflammation
MeSH Terms: conditions — Hypertension; Inflammation | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- abatacept (Active Comparator): Subjects randomized to abatacept weighing 60 to 100 kg will receive 750 mg, and those >100 kg will receive 1000 mg abatacept by intravenous infusion at 0 [randomization], 2, and 4 weeks and then every 4 weeks thereafter for a total of 24 weeks.
  All subjects will be treated with chlorthalidone 25 mg/day, lisinopril 20 mg/day [Patients with a history of adverse reaction to lisinopril will be treated with losartan 50 mg/day], amlodipine 5 mg/day and spironolactone 25 mg bid as standardized treatment of hypertension prior to randomization and throughout the active treatment phase.
  Interventions: Drug: Abatacept
- placebo (Placebo Comparator): Subjects randomized to placebo will receive 100 ml normal saline by intravenous infusion at 0 [randomization], 2, and 4 weeks and then every 4 weeks thereafter for a total of 24 weeks.
  All subjects will be treated with chlorthalidone 25 mg/day, lisinopril 20 mg/day [Patients with a history of adverse reaction to lisinopril will be treated with losartan 50 mg/day], amlodipine 5 mg/day and spironolactone 25 mg bid as standardized treatment of hypertension prior to randomization and throughout the active treatment phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abatacept — All subjects will be treated with chlorthalidone 25 mg/day, lisinopril 20 mg/day [Patients with a history of adverse reaction to lisinopril will be treated with losartan 50 mg/day], amlodipine 5 mg/day and spironolactone 25 mg bid as standardized treatment of hypertension prior to randomization and throughout the active treatment phase.
  Other Names: Orencia
  Arms: abatacept
Drug: Placebo — All subjects will be treated with chlorthalidone 25 mg/day, lisinopril 20 mg/day [Patients with a history of adverse reaction to lisinopril will be treated with losartan 50 mg/day], amlodipine 5 mg/day and spironolactone 25 mg bid as standardized treatment of hypertension prior to randomization and throughout the active treatment phase.
  Arms: placebo

SUMMARY:
The purpose of this study is to test whether abatacept, a drug approved by the Food and Drug Administration to treat rheumatoid arthritis, may help blood pressure medications to work better. This will be studied in people with high blood pressure that is not well controlled on three or more blood pressure medications, the condition also known as resistant hypertension. We expect to show that adding abatacept therapy to standardized treatment of resistant hypertension will result in a greater decrease in blood pressure at 24 weeks compared to treatment with placebo and conventional blood pressure treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 65 years of age with hypertension, treated with three or more anti-hypertensive drugs, one being a diuretic, and
* having a systolic blood pressure >150 mmHg in the clinic and daytime average >150 mmHg on ambulatory blood pressure monitoring

Exclusion Criteria:

* Medical history of secondary cause of hypertension, severe obesity (BMI >35), severe psychiatric disorders, cancer in the last 5 years other than nonmelanoma skin cell cancers, herpes zoster or cytomegalovirus that resolved less than 2 months before
* Inability to return for abatacept treatment and follow-up for 24 weeks.
* Inability to understand or complete study-related assessments.
* Current abuse of drugs or alcohol.
* Receipt of any live vaccines within 3 months of the anticipated first dose of study medication.
* Evidence of active or latent bacterial or viral infections at the time of potential enrollment, including human immunodeficiency virus (HIV)
* Risk for tuberculosis
* Abnormal laboratory values including positive hepatitis B surface antigen, hemoglobin < 8.5 g/dL, white blood cell count < 3000/mm3, platelets < 100,000/mm3, creatinine > 2.5 times the upper limit of normal (ULN), alanine aminotransferase or aspartate aminotransferase > 2 times the ULN.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G Harrison, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was consented. The study terminated before the participant was randomized. No participants received treatment.
Period: Overall Study
Arm/Group | Consented Patients
Started | 1
Completed | 0
Not Completed | 1
Not completed — study stopped prior to randomization | 1

BASELINE CHARACTERISTICS:
Groups:
- Consented Patients: No patients received treatment prior to study termination
Arm/Group | Consented Patients
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure From Randomization to End of Treatment
Description: Ambulatory blood pressure monitoring will be used at the end of the 4 weeks standardized treatment and at the end of 6 months randomized treatment with abatacept or placebo. The change in systolic blood pressure from these 2 recordings will be the primary endpoint.
Time Frame: 6 months
Population: No patients received treatment prior to study termination
Arm/Group | Consented Patients
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Blood Pressure
Description: Changes in the rate of change of blood pressure estimated by automated in office cuff measurements and ambulatory blood pressure at 12 weeks after randomization
Time Frame: 6 months
Population: No patients received treatment prior to study termination.
Arm/Group | Consented Patients
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Brachial Artery Reactivity
Description: change in brachial artery reactivity measured at randomization and after 24 weeks of treatment
Time Frame: 6 months
Population: No patients received treatment prior to study termination
Arm/Group | Consented Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Inflammatory Markers
Description: changes in plasma and T cell markers of activation and T cell cytokine production from randomization to end of 24 weeks of treatment
Time Frame: 6 months
Population: No patients received treatment prior to study termination
Arm/Group | Consented Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: One participant was consented. The study terminated before the participant was randomized. No participants received treatment.
Arm/Group | Consented Patients
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
No patients received treatment prior to study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No